CLINICAL TRIAL: NCT00737789
Title: Multicentre, Controlled, Randomised, Investigator-Blinded, Comparative Study of Oral Mesalazine 4g Once Daily Versus Mesalazine 4g in Two Divided Doses in Patients With Active Ulcerative Colitis.
Brief Title: Mesalazine 4g Once Daily Versus 4g in Two Divided Doses in Active Ulcerative Colitis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pentasa FE999907 CS06; EudractCT No 2008-000045-59
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mesalazine once/day (Experimental): Participants received 4g oral Mesalazine once a day (2 sachets of prolonged release granules) for 8 weeks during the induction period. In addition, participants received a liquid enema of 1g Mesalazine once a day at bedtime for the first 4 weeks. Participants who were in remission at Week 8 received oral mesalazine 2g once daily (1 sachet/day) for an additional 4 weeks (maintenance period).
  Interventions: Drug: Mesalazine slow-release granules; Drug: Mesalazine liquid enema
- Mesalazine twice/day (Active Comparator): Participants received oral mesalazine 4 g per day in two divided doses (1 sachet prolonged release granules twice a day) for 8 weeks during the induction period. In addition, participants received a liquid enema of 1g Mesalazine once a day at bedtime for the first 4 weeks. Participants who were in remission at Week 8 received oral Mesalazine 2g (one sachet) once a day for an additional 4 weeks (maintenance period).
  Interventions: Drug: Mesalazine slow-release granules; Drug: Mesalazine liquid enema

INTERVENTIONS:
Drug: Mesalazine slow-release granules — Mesalazine 2g Sachet prolonged release granules, administered orally.
  Other Names: Pentasa
Drug: Mesalazine liquid enema — 1g mesalazine liquid enema, administered topically once a day in the evening.

SUMMARY:
The purpose of this study was to demonstrate that mesalazine 4g orally per day once daily (QD) is non-inferior to the reference regimen, mesalazine 4g per day in two divided doses (BID) (2g x 2 per day), in patients with active ulcerative colitis (UC) treated for 8 weeks, in terms of remission evaluated with the Ulcerative Colitis Disease Activity Index (UC-DAI) score and defined as less than or equal to 1. Both groups (4g QD and 2gx2) received an enema containing 1g of mesalazine at bedtime during the initial 4 weeks.

Participants in remission at week 8 received an additional 4 weeks of maintenance therapy with 2g oral mesalazine once a day. Participants who did not achieve remission at Week 8 completed the study at week 8.

DETAILED DESCRIPTION:
A key element in therapeutic response in UC is treatment compliance. In daily practice, compliance of UC patients with 5-Amino Salicylic Acid (5-ASA) treatment appears mediocre, particularly in maintenance therapy. Poor or non-existent compliance affects not only treatment response but also disease progression.

An inverse relationship has been found between the number of daily doses prescribed and treatment compliance. Thus, reduction to a single daily dose of mesalazine is a major factor likely to significantly increase treatment compliance.

Reducing the dosing rate to a single daily dose for 8 weeks constitutes a simple method of improving treatment compliance but it is necessary to demonstrate at least equivalent efficacy compared to the twice daily dosing which is the reference regimen. This study was designed to show that mesalazine 4g once daily is at least as effective as mesalazine 4g in two divided doses per day in patients with mild to moderate ulcerative colitis after 8 weeks of treatment with a better compliance. To improve remission, both groups received an enema during the first 4 weeks, as usually done in current practice.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included if they comply with the following inclusion criteria determined at baseline, prior to first drug administration:

* Aged over 18 years.
* Newly diagnosed or relapsing mild to moderate ulcerative colitis with disease extension beyond rectum (of at least 12-18 cm from the anorectal junction). All patients must have had at least one total colonoscopy in their disease history (within the previous 5 years).
* Disease activity will be assessed on the 15 days before inclusion and according to ulcerative colitis disease activity index (UC-DAI) score. The UC-DAI score will be from 3 to 8 (mild: 3-5 or moderate: 6-8).
* Men or non pregnant women.
* Women with childbearing potential must be using a contraceptive method judged effective by the investigator.
* Oral maintenance treatment with azathioprine or 6-mercaptopurine (taken for at least 6 months at stable dose and continued at the same dose throughout the study) is permitted.
* Informed consent given.

Exclusion Criteria:

The patients will not be included in the study if one of the following exclusion criteria is fulfilled at baseline, prior to first drug administration:

* Proctitis (less than 12-18 cm from the anorectal junction).
* Previous colonic surgery.
* Previously failed to respond to steroids within the previous year.
* Non-response to rectal 5-Amino Salicylic Acid (5-ASA) therapy or to oral 5-ASA therapy at a dose > 3g/day for induction of remission within the previous year.
* Current relapse lasting more than 6 weeks (for patient recently diagnosed the period of 6 weeks runs from the endoscopic diagnosis)(from what patient says).
* Severe/fulminant ulcerative colitis.
* Evidence of other forms of inflammatory bowel disease or infectious disease.
* Allergy to aspirin or salicylate derivatives.
* The following treatment will be forbidden during the study (if present at selection, a wash-out will be necessary):
* Loperamide and other antidiarrheal agents, mucilages, antibiotics: 1 week wash-out.
* Oral steroids: 4 weeks wash-out.
* Rectal steroids: 2 weeks wash-out
* Repeated treatment (> 3days of use) of non steroidal anti-inflammatory drugs (NSAID) oral or rectal route: 1 week wash-out (aspirin ≤ 325 mg/day used for cardioprotection is allowed).
* Sulfasalazine > 4g/day or mesalazine or 4-ASA at a higher dose than what is permitted in the local formulary or standard care for maintenance treatment: 4 weeks wash-out
* Immunomodulating/suppressing drugs: 3 month for wash out (except for patients maintained on azathioprine or 6-mercaptopurine -see above).
* Known significant hepatic or renal function abnormalities.
* Moderate/severe abnormal renal, hepatic or blood count tests defined as: creatinine plasma value > 1.5 x Upper Limit of Normal (ULN) or white blood cells < 3500/mm˄3 or > 15000/mm˄3 or Platelets < 100000/mm˄3 or > 800000/mm˄3 or aspartate aminotransferase/alanine Aminotransferase (ASAT/ALAT) > 3 x ULN or Gamma glutamyl transpeptidase (GGT)/Alkaline Phosphatase's > 3 x ULN (Primary Sclerosing Cholangitis is not an exclusion criteria).
* History or physical examination findings indicative of active alcohol or drug abuse,
* Pregnancy or breast-feeding,
* History of disease, including mental/emotional disorder, that might interfere with their participation in the study,
* Participation in another clinical study in the last 3 months.
* Inability to comply with the protocol requirements.
* Inability to fill in the diary cards.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2008-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Primary efficacy criterion: remission after 8 weeks of treatment, defined on the basis of the UC-DAI score less than or equal to 1 | 12 weeks

SECONDARY OUTCOMES:
Compliance | Week 8
Clinical remission | At week 4, week 8 and week 12
Treatment failure is defined as need of other treatment (ie steroids, immunosuppressive or immunomodulating drugs) than those allowed by the protocol, as judged by investigator. Treatment failure will be counted as non-remission. | At week 4 and week 8
Clinical variables (stool frequency and bloody stools) | At week 4, 8 and 12 separately
Time to remission according to patient's diary (normal stool frequency and cessation of bleeding) | At week 4 and week 8
Time to cessation of bleeding | At week 4, week 8 and week 12
Improvement - based on UC-DAI score | At week 4 and 8
Endoscopic assessment | At week 0 and week 8
Safety | At week 0, week 4, week 8 and week 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (66):
- Belgium (6):
  - O.L.Vrouwziekenhuis Campus Aalst, Aalst
  - C.H.U. Saint-Pierre, Brussels
  - Saint Luc University Hospital, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - U.Z. Antwerpen, Edegem
  - University Hospital Gasthuisberg, Leuven
- France (50):
  - Clinique Esquirol-St Hilaire, Agen
  - Investigational site, Albi
  - Investigational site, Amiens
  - Centre Hospitalier Avignon, Avignon
  - Centre Hospitalier Bethune, Béthune
  - Investigational site, Bourgoin
  - Investigational site, Brest
  - Clinique Jean-Villar, Bruges
  - Clinique Saint Martin - 18 rue Rocquemonts, Caen
  - Clinique Saint Martin, Caen
  - Investigational site, Caluire-et-Cuire
  - Investigational site, Carcassonne
  - Clinique du Parc, Castelnau-le-Lez
  - Investigational site, Chambray-lès-Tours
  - Centre Médical République, Clermont-Ferrand
  - Investigational site, Clichy
  - Clinique des Cèdres, Cornebarrieu
  - Centre Hospitalier Intercommunal, Créteil
  - Investigational site, Dunkirk
  - Centre Hospitalier Universitaire Albert MICHALON, Grenoble
  - Investigational site, Grenoble
  - Investigational site, Hazebroucq
  - Investigational site, Irigny
  - Investigational site, Istres
  - Centre Hospitalier Lagny, Lagny
  - Investigational site, Le Mans
  - Investigational site - 23 bis, place Sébastol, Lille
  - Investigational site - 60 rue Jean Bart, Lille
  - Clinique de la Sauvegarde, Lyon
  - Investigational site - 186 avenue de la Rose, Marseille
  - Investigational site - 23 Cours Gouffé, Marseille
  - Investigational site, Miramas
  - CH Le raincy-Montfermeil, Montfermeil
  - Investigational site, Nancy
  - Hôpital L'Archet 2, Nice
  - Investigational site - 127 boulevard St Germain, Paris
  - Investigational site - 72 rue Archeveau, Paris
  - Investigational site - 91 rue Caulaincourt, Paris
  - Investigational site, Perpignan
  - Clinique Saint Martin, Pessac
  - Hôpital de Lyon Sud, Pierre-Bénite
  - Investigational site, Reims
  - Centre Hospitalier Privé, Saint-Grégoire
  - Investigational site - 140 avenue Lwoff, Saint-Priest
  - Investigational site, Saint-Quentin
  - Investigational site, Strasbourg
  - Clinique Saint Jean Languedoc - 20 route de Revel, Toulouse
  - Clinique Saint Jean-Languedoc, Toulouse
  - Centre FUTURA MEDICA, Verquigneul
  - Groupe Hospitalier les Portes du Sud, Vénissieux
- Netherlands (7):
  - Kennemer Gasthuis, loc. EG, Haarlem
  - Streekziekenhuis Midden Twente, Hengelo
  - IJsselmeer Ziekenhuis Loc. Lelystad, Poli MDL, Lelystad
  - Mumc / Azm, Maastricht
  - Haga Ziekenhuis, loc.Rode Kruis, The Hague
  - TweeSteden Ziekenhuis, Tilburg
  - Isala Klinieken, loc. Sophia, Zwolle
- United Kingdom (3):
  - Bristol Royal Infirmary, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Royal Victoria Infirmary, Newcastle

REFERENCES:
- [Derived] Flourie B, Hagege H, Tucat G, Maetz D, Hebuterne X, Kuyvenhoven JP, Tan TG, Pierik MJ, Masclee AA, Dewit O, Probert CS, Aoucheta D; MOTUS study investigators. Randomised clinical trial: once- vs. twice-daily prolonged-release mesalazine for active ulcerative colitis. Aliment Pharmacol Ther. 2013 Apr;37(8):767-75. doi: 10.1111/apt.12266. Epub 2013 Mar 4. PMID 23451806